CLINICAL TRIAL: NCT05612321
Title: All-fours Position vs Traditional Position in Women Undergoing Vacuum-assisted Delivery: the VaDe-4 Randomized Controlled Trial
Brief Title: Vacuum Delivery in All-fours Position vs Traditional Position
Acronym: VaDe-4
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ospedale degli Infermi di Biella (Other)
Responsible Party: Principal Investigator, Bianca Masturzo, Head of Department of Gynaecology and Obstetrics, Ospedale degli Infermi di Biella
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VaDe-4/2022
Record Dates: First submitted 2022-10-19; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Prolonged Second Stage of Labor; Prolonged Second Stage of Labor Due to Poor Maternal Effort
Keywords: Vacuum-assisted vaginal delivery; All-fours position; Arrest of descent; Operative vaginal delivery
MeSH Terms: conditions — Cephalopelvic Disproportion

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomized open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Traditional supine position (Active Comparator): Participants enrolled in the Control Group undergo vacuum-assisted delivery in traditional supine position (supine with 90 degrees bended legs on footrests)
  Interventions: Device: Vacuum application
- All-fours position (Experimental): Participants enrolled in Experimental Group experience vacuum application in all-fours position.
  Interventions: Device: Vacuum application

INTERVENTIONS:
Device: Vacuum application — vacuum-assisted delivery

SUMMARY:
The aim of the study is to investigate the safety, clinical efficacy and the maternal/neonatal outcomes of vacuum application in all-fours position compared with supine traditional position, in women undergoing vacuum-assisted delivery during the second stage of labor.

The main question it aims to answer are:

* Does the rate of failure of vacuum delivery, measured as number of cup detachments and the need of emergency caesarean section is lower if vacuum delivery is performed on a woman in all-fours position?
* Do maternal and fetal outcomes are better in case vacuum delivery in all-fours position?

Participants will be randomly enrolled at the admission in two different groups, Control and Experimental Group, and in case of need for vacuum-assisted vaginal delivery; women belonging to Control Group will undergo vacuum-assisted delivery in traditional supine position, while women in Experimental Group will experience vacuum application in all-fours position.

Researchers will compare the Group A, composed by women who undergo vacuum-delivery in traditional supine position, with Group B, in which women are in "all-fours" position, to see if hands-and-knees position provides better outcomes.

DETAILED DESCRIPTION:
In the last decades, a decrease in operative vaginal delivery (OVD) rates occurred, resulting in increase of caesarean sections (CS) during the second stage of labor. This attitude reflects Clinicians' worries about operative vaginal delivery morbidity, together with a consequent loss of clinical skills in this practice. However, vacuum delivery - when correctly performed - requires less analgesia and gives women higher chances to have a spontaneous vaginal birth in the following pregnancy, whereas emergency C-section is burdened by different maternal and fetal complications. Moreover, should fetal compromise be occurring, time to start the procedure is longer for CS than for vacuum application. Due to the whole of these reasons, operative vaginal delivery is included in the main international guidelines as the best option for the mother and baby, in case of arrest/delay of fetal head descent during second stage of labor, with fetal head at mid/low-pelvic station.

Although women in labor are usually asked to choose the position they prefer and to change position frequently to facilitate the alignment of the fetal head with the birth canal, the vacuum cup is usually applied to a woman lying in the "traditional" gynecological supine position.

Despite several demonstrated advantages, fewer women choose non-recumbent positions, and among them, the so-called "all-fours position" (or "hands-and-knees") which has the higher evidence of benefit. In all-fours, the woman is on her knees, leaning on her hands, with abdomen suspended and hips at right angles to the floor or bed. As demonstrated in different studies, the main advantage given by this posture is the increase of all posterior diameters of the pelvis. This finding implies not only an easier descent of the fetal head, helped by gravity, but also a wider space where fetal head could rotate in case of occiput posterior position, preventing fetal malposition. Additionally, this position lets the sacrum to have more posterior mobility (contra-nutation movement) furtherly widening the outlet no more constricted by the standing surface and reducing sacral pain due to bed-contact. Moreover, as the burden of trunk's weight on the sacrum is decreased in all-fours, women consider the hands-and-knees position a pain-relieving postural choice, especially during the first stage of labor. Regarding maternal outcomes, a recent large randomized controlled trial, involving 1400 women, demonstrated a lower incidence of second-degree perineal lacerations, episiotomy and perineal swelling in hands-and-knees position, and a lower risk of emergency CS, compared to other birth positions.

In the all-fours position, the vaginal space between the fetal head and the vaginal ostium is not influenced by body weight, resulting wider, visible, and easily explorable. Moreover, the risk of vacuum cup sliding is lower because the upward traction is allotted a wider space.

The widening of birth canal obtained with this technique has several, beneficial implications. First, the risk of vaginal tear is lower, since there is no redundant vaginal tissue that could be trapped inside the cup. Second, a wider space allows to constantly maintain the vacuum wire perpendicular to the cup, thus determining a lower risk of detachment, subsequent fetal scalp damage and cephalohematoma (e.g., in presence of caput succedaneum).

Also, this position allows a better propulsive pushing, thanks to a more efficient Valsalva maneuver, thus enabling the Clinician not to exert excessive traction on the fetal head.

Since OVD has a known increased risk of shoulder dystocia, adopting the all-fours position should be beneficial in preventing this fearsome complication, consistent with the point that the hands-and-knees posture is required to perform the Gaskin maneuver, a rescue procedure that easily releases the trapped shoulder by taking advantage of the greater posterior pelvic space in this position.

A potential disadvantage might be the inability of the woman to keep this position for longer than 10-15 minutes. Although OVD duration is routinely much shorter, it is of course mandatory that the timing of OVD performance be carefully monitored.

The investigators recently suggested the implementation of all-fours position in case of operative vaginal delivery and we published a video-simulation of vacuum application on a mannequin. At this time, no other prospective study so far assessed a putative effectiveness of an alternative positioning strategy during OVD for women with arrest of fetal head progression during the second stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* women
* singleton
* cephalic presentation
* term pregnancy
* second stage of labor
* failure to progress
* maternal weariness
* need for operative vaginal delivery by vacuum extraction

Exclusion Criteria:

* enrollment refusal
* absence of consent
* contraindication to operative vaginal delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study requires the enrollement of only female participants as it refers to delivery.
Enrollment: 250 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Vacuum detachments | Day 0
  Vacuum detachments (Yes/No)
Rate of Emergency C-Section | Day 0
  Emergency C-section (Yes/No)

SECONDARY OUTCOMES:
Perineal tears | Day 1
  Perineal tears (1st-3rd grade) (Yes/No and Grade: 1st/2nd/3rd grade)
Obstetric anal sphincter injuries (OASIS) | Day 1
  Obstetric anal sphincter injuries (OASIS, 4th grade) (Yes/No)
Episiotomy | Day 1
  Episiotomy (Yes/No)
Blood loss | Day 1
  Maternal blood loss (ml)
Postpartum haemorrhage | Day 1
  Postpartum haemorrhage defined as a blood loss of >1000milliliters (Yes/No)
Necessity of Blood Transfusions | Day 3
  Blood Transfusions (Yes/no and n. bagged blood infused)
Maternal infections | Day 3
  Maternal infections (endometritis, sepsis, hyperpyrexia) (Yes/No)
Length of Hospital Stay | Day 30
  Length of Hospital Stay (n. of days of hospitalization)
Patient Satisfaction | Day 30
  Short-form patient satisfaction questionnaire (PSQ-18) (18 and 90 are the minimum and maximum values, and higher scores mean a higher patient satisfaction).
APGAR score | Day 0
  APGAR score at 1 and 5 minutes (0-10)
Neonatal acidosis | Day 0
  pH < 7.10 at birth (Yes/No)
Neonatal hypoglycaemia | Day 1
  Neonatal Serum Glucose < 45 mg/dL (< 2.5 mmol/L) (Yes/No)
Neonatal cephalohematoma | Day 1
  Neonatal cephalohematoma (Yes/No)
Neonatal scalp damages | Day 1
  Neonatal scalp damages (Yes/No)
Shoulder Dystocia | Day 0
  Shoulder Dystocia (Yes/No)
Admission to Neonatal Intensive Care Unit (NICU) | Day 30
  Admission to Neonatal Intensive Care Unit (NICU) (Yes/No)
Need for Oxygen Supplementation | Day 30
  Neonatal need for supplementary oxygen (yes/no) and days of use (days)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Masturzo, Md, PhD, Principal Investigator — Ospedale degli Infermi di Biella

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, CSR
Time Frame: At the end of the study, for 6 months from the 1st Jan 2024 to 1st July 2024
Access Criteria: Participants centers

REFERENCES:
- [Result] Merriam AA, Ananth CV, Wright JD, Siddiq Z, D'Alton ME, Friedman AM. Trends in operative vaginal delivery, 2005-2013: a population-based study. BJOG. 2017 Aug;124(9):1365-1372. doi: 10.1111/1471-0528.14553. Epub 2017 Feb 25. PMID 28236337
- [Result] Spencer C, Murphy D, Bewley S. Caesarean delivery in the second stage of labour. BMJ. 2006 Sep 23;333(7569):613-4. doi: 10.1136/bmj.38971.466979.DE. No abstract available. PMID 16990297
- [Result] Guo C, Ma W, Fan D, Ma Y, Liu L. Non spontaneous vaginal delivery was associated with lower probability of subsequent fertility. Eur J Obstet Gynecol Reprod Biol. 2020 May;248:30-36. doi: 10.1016/j.ejogrb.2020.03.009. Epub 2020 Mar 7. PMID 32172023
- [Result] Operative Vaginal Birth: ACOG Practice Bulletin, Number 219. Obstet Gynecol. 2020 Apr;135(4):e149-e159. doi: 10.1097/AOG.0000000000003764. PMID 32217976
- [Result] RANZCOG. The Women's Health Committee. The Royal Australian and New Zealand College of Obstetricians and Gynaecologists. Instrumental vaginal birth; March 2016.
- [Result] Hobson S, Cassell K, Windrim R, Cargill Y. No. 381-Assisted Vaginal Birth. J Obstet Gynaecol Can. 2019 Jun;41(6):870-882. doi: 10.1016/j.jogc.2018.10.020. PMID 31126436
- [Result] Murphy DJ, Strachan BK, Bahl R; Royal College of Obstetricians and Gynaecologists. Assisted Vaginal Birth: Green-top Guideline No. 26. BJOG. 2020 Aug;127(9):e70-e112. doi: 10.1111/1471-0528.16092. Epub 2020 Apr 28. No abstract available. PMID 32346983
- [Result] Stremler R, Hodnett E, Petryshen P, Stevens B, Weston J, Willan AR. Randomized controlled trial of hands-and-knees positioning for occipitoposterior position in labor. Birth. 2005 Dec;32(4):243-51. doi: 10.1111/j.0730-7659.2005.00382.x. PMID 16336365
- [Result] Siccardi M, Valle C, Di Matteo F. Dynamic External Pelvimetry Test in Third Trimester Pregnant Women: Shifting Positions Affect Pelvic Biomechanics and Create More Room in Obstetric Diameters. Cureus. 2021 Mar 1;13(3):e13631. doi: 10.7759/cureus.13631. PMID 33816030
- [Result] Michel SC, Rake A, Treiber K, Seifert B, Chaoui R, Huch R, Marincek B, Kubik-Huch RA. MR obstetric pelvimetry: effect of birthing position on pelvic bony dimensions. AJR Am J Roentgenol. 2002 Oct;179(4):1063-7. doi: 10.2214/ajr.179.4.1791063. PMID 12239066
- [Result] Hemmerich A, Bandrowska T, Dumas GA. The effects of squatting while pregnant on pelvic dimensions: A computational simulation to understand childbirth. J Biomech. 2019 Apr 18;87:64-74. doi: 10.1016/j.jbiomech.2019.02.017. Epub 2019 Feb 27. PMID 30851977
- [Result] Zhang H, Huang S, Guo X, Zhao N, Lu Y, Chen M, Li Y, Wu J, Huang L, Ma F, Yang Y, Zhang X, Zhou X, Guo R, Cai W. A randomised controlled trial in comparing maternal and neonatal outcomes between hands-and-knees delivery position and supine position in China. Midwifery. 2017 Jul;50:117-124. doi: 10.1016/j.midw.2017.03.022. Epub 2017 Mar 31. PMID 28414983
- [Result] Bothou A, Apostolidi DM, Tsikouras P, Iatrakis G, Sarella A, Iatrakis D, Peitsidis P, Gerente A, Anthoulaki X, Nikolettos N, Zervoudis S. Overview of techniques to manage shoulder dystocia during vaginal birth. Eur J Midwifery. 2021 Oct 20;5:48. doi: 10.18332/ejm/142097. eCollection 2021. PMID 34723155
- [Result] Masturzo B, Delogu G, Germano C, Ghi T, Rizzo G, Puppo A, Attini R, Revelli A, Manzoni P. Vacuum delivery in all-fours position: is it a valuable, brand-new option? Am J Obstet Gynecol MFM. 2022 Nov;4(6):100691. doi: 10.1016/j.ajogmf.2022.100691. Epub 2022 Jul 16. PMID 35843544